CLINICAL TRIAL: NCT06759623
Title: Assessment of Pulmonary Function in Relation to the Anesthetic Used in Patients Undergoing Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radosław Owczuk, Prof. dr hab., Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KO_bariatria
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General anesthesia with desflurane (Experimental): Patients undergoing anesthesia for bariatric surgery with desflurane as a volatile agent.
  Interventions: Drug: Different drug type for conduction of general anesthesia
- General anesthesia with sevoflurane (Experimental): Patients undergoing anesthesia for bariatric surgery with sevoflurane as a volatile agent.
  Interventions: Drug: Different drug type for conduction of general anesthesia

INTERVENTIONS:
Drug: Different drug type for conduction of general anesthesia — Patients will be randomly divided into two groups: patients for whom general anesthesia will be performed with sevoflurane and patients for whom general anesthesia will be performed with desflurane.

SUMMARY:
It is known that more or less pronounced impairment of pulmonary function occurs after anesthesia. It has been demonstrated in the postoperative period in both patients undergoing general and regional anesthesia, in patients after intra-abdominal and superficial procedures, in overweight and normal-weight patients. It has also been shown that when general anesthesia is performed with the inhalation anesthetic sevoflurane, there is a slightly smaller reduction in lung function parameters than when only intravenous anesthetics are used.

The purpose of this study is to evaluate lung function before induction and after awakening from general anesthesia depending on the inhalational anesthetic used in obese patients undergoing bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* Obese patients qualified for bariatric surgery.

Exclusion Criteria:

* Patients who have absolute contraindications to spirometry testing, i.e:

  * with aneurysms of the aorta or cerebral arteries threatening to rupture, after recent vascular surgery
  * with increased intracranial pressure, after recent intracranial bleeding or head surgery within the cranial cavity
  * after acute conditions within 6 months prior to surgery such as stroke, myocardial infarction, unstable angina, pneumothorax
  * with uncontrolled hypertension
  * after recent eye surgery or a history of retinal detachment
  * with hemoptysis of unknown etiology. And patients unable to perform spirometry testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-08 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate (HR) | Continuously during whole duration of anesthesia
  HR will be measured by ecg in beat per minute
Pulse oximetry (SpO2) | Continuously during whole duration of anesthesia
  SpO2 will be measured by light spectrometry percutaneous sensor in %
End tidal CO2 (etCO2) | Continuously during whole duration of anesthesia
  etCO2 will be measured by capnography with infrared radiation sensor in mmHg. Sensor will be attached to breathing circuit.
Minimum alveolar concentration (MAC) | Continuously during whole duration of anesthesia
  MAC will be measured based on exhaled anesthetic gas concentration in absolute numbers
Bispectral index (BIS) | Continuously during whole duration of anesthesia
  BIS will be measured with Covidien BIS monitoring system in absolute numbers
Train of for (TOF) | Every 2.5 minutes during whole duration of anesthesia
  TOF will be measured in absolute numbers
Non invasive blood pressure (NIBP) | Every 5 minutes during whole duration of anesthesia
  NIBP will be measured with oscillometric method in mmHG
Forced vital capacity (FVC) | 3 months before the surgery and 10 and 30 minutes after the emergence from general anesthesia
  FVC will be measured with spirometry
Volume that has been exhaled at the end of the first second of forced expiration (FEV1) | 3 months before the surgery and 10 and 30 minutes after the emergence from general anesthesia
  FEV1 will be measured with spirometry
Mid-expiratory flow; the rates at 25% FVC (MEF25) | 3 months before the surgery and 10 and 30 minutes after the emergence from general anesthesia
  MEF25 will be measured with spirometry
Mid-expiratory flow; the rates at 25% FVC (MEF50) | 3 months before the surgery and 10 and 30 minutes after the emergence from general anesthesia
  MEF50 will be measured with spirometry
Peak expiratory flow (PEF) | 3 months before the surgery and 10 and 30 minutes after the emergence from general anesthesia
  PEF will be measured with spirometry
Respiratory input impedance (Zrs) | 3 months before the surgery and 10 and 30 minutes after the emergence from general anesthesia
  Zrs will be measured with impulsed oscillometry
Resistive component (Rrs) | 3 months before the surgery and 10 and 30 minutes after the emergence from general anesthesia
  Rrs will be measured with impulsed oscillometry
Reactive component (Xrs) | 3 months before the surgery and 10 and 30 minutes after the emergence from general anesthesia
  Xrs will be measured with impulsed oscillometry
Resonant frequency (Fres) | 3 months before the surgery and 10 and 30 minutes after the emergence from general anesthesia
  Fres will be measured with impulsed oscillometry
Area of reactance (Ax) | 3 months before the surgery and 10 and 30 minutes after the emergence from general anesthesia
  Ax will be measured with impulsed oscillometry

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No